CLINICAL TRIAL: NCT04023903
Title: A Clinical Pharmacology Study of RTA 402 (Investigation of the Effect of Food on the Pharmacokinetics of RTA 402 Capsules in Japanese Healthy Adults and Comparison of the Pharmacokinetics With Those in Caucasian Healthy Adults)
Brief Title: A Clinical Pharmacology Study of Bardoxolone Methyl in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RTA 402-009
Record Dates: First submitted 2019-07-16; First posted 2019-07-18 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Healthy Subject
Keywords: Bardoxolone Methyl; Healthy subject; Food effect
MeSH Terms: interventions — bardoxolone methyl

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RTA 402 5mg 3cap at fasting (Experimental)
  Interventions: Drug: Bardoxolone methyl
- RTA 402 5mg 3cap after meal (Experimental)
  Interventions: Drug: Bardoxolone methyl

INTERVENTIONS:
Drug: Bardoxolone methyl — Bardoxolone methyl 5 mg capsules
  Other Names: RTA 402
  Arms: RTA 402 5mg 3cap at fasting
Drug: Bardoxolone methyl — Bardoxolone methyl 5 mg capsules
  Other Names: RTA 402
  Arms: RTA 402 5mg 3cap after meal

SUMMARY:
Food effect part:

To investigate the effect of food on the pharmacokinetics of RTA 402 and evaluate the safety of RTA 402 in Japanese healthy male adults, using the capsule formulations.

Caucasian subject part:

To investigate the pharmacokinetics of a single dose of RTA 402 administered in the fasted state and compare the pharmacokinetics with those observed in Japanese healthy male adults in the food effect part

ELIGIBILITY:
Inclusion Criteria:

1) Written voluntary informed consent to participate in the study; 2) [Food Effect Part] Japanese men 20 to <40 years of age at informed consent; [Caucasian Subject Part] Caucasian men 20 to <40 years of age at informed consent; 3) BMI 18.5 kg/m2 to <25.0 kg/m2 at screening

Exclusion Criteria:

1. Presence of any disease requiring treatment;
2. History of heart failure (e.g., history of diagnosis of congestive heart failure categorized as Class III or IV of the New York Heart Association (NYHA) Functional Classification or history of hospitalization due to heart failure);
3. Alcoholism or drug addiction, or any positive result on drug abuse testing;
4. History of or current drug allergy;
5. Any positive result on infectious disease testing. Individuals who are positive for active antibodies produced by hepatitis B vaccination and are not infected with hepatitis B virus at screening can be enrolled in the study;

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 36 (Actual)
Dates: Start 2019-04-04 (Actual); Primary Completion 2019-06-14 (Actual); Study Completion 2019-06-14 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours
AUC0-t | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours

SECONDARY OUTCOMES:
tmax | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours
AUC0-∞ | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours
t1/2 | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours
MRT | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours
kel | Pre-dose, 0.5, 1, 2, 4, 6, 8, 10, 12, 24, 30, 36, 48, 60, 72, 96 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Corporation Heishinkai OPHAC Hospital, Osaka, Japan

IPD SHARING:
Plan to Share IPD: Undecided